CLINICAL TRIAL: NCT05281484
Title: Two Intermediate Expanded Access Protocols for Amyotrophic Lateral Sclerosis With CNM-Au8. CNMAu8.EAP01 and CNM.EAP02
Brief Title: Two Intermediate Expanded Access Protocols (EAP) CNMAu8.EAP01 and CNMAu8.EAP02 for ALS
Status: Available | Type: Expanded Access
Sponsor: Clene Nanomedicine (Industry)
Responsible Party: Sponsor
Other Study IDs: CNMAu8.EAP 01 & 02
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Expanded access; ALS; Amyotrophic Lateral Sclerosis; CNM Au8; Au8
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: CNM-Au8 — CNM-Au8 is an aqueous suspension of clean surfaced faceted nanocrystals consisting of gold atoms self-organized into crystals of various geometrical shapes (hexagonal bi-pyramid, pentagonal bipyramid, tetrahedron, decahedron, planar spheroids).
  Highly pure elemental Au nanocrystals are suspended in USP purified deionized water buffered with 0.546 mg/mL (6.5 mM) sodium bicarbonate (NaHCO3) nominally concentrated to up to 0.5 mg/mL (500 ppm).
  Other Names: Nanocrystalline gold

SUMMARY:
The primary objective of the intermediate expanded access protocol is to provide access to the investigational product, CNM-Au8, to up to 300 people living with ALS (pALS).

No formal clinical hypotheses are being evaluated with concurrent controls.

Secondary objectives include assessment of the safety of CNM-Au8 treatment in pALS. Safety will be assessed through the frequency of serious adverse events (SAEs), treatment-emergent adverse events (TEAEs) assessed as 'severe', discontinuations due to TEAEs, and laboratory abnormalities assessed as clinically significant during routine clinical monitoring (as applicable).

DETAILED DESCRIPTION:
This is a multi-center intermediate expanded access program to provide access to the investigational product, CNM-Au8, up to 300 participants diagnosed with ALS.

The safety of CNM-Au8 treatment in ALS participants will be evaluated. Visits will occur at a clinic or remotely via telephone or video-visit. Visits may be conducted remotely due to COVID-19-related pandemic concerns, or if due to ALS disease progression.

Participants who meet the inclusion criteria and none of the exclusionary criteria may be enrolled into the EAP.

There will be three study periods:

1. A treatment period of forty-eight (48) weeks (Treatment Period 1);
2. Additional optional follow-on treatment period(s) of up to forty-eight (48) weeks duration may be added at the discretion of the Sponsor and Site Investigator (e.g., Treatment Period 2, Treatment Period 3);
3. A four (4) week safety follow-up period (End-of-Study [EOS]Assessment).

All participants will receive open-label oral treatment daily up to 48 weeks during Treatment Period 1. Additional 48-week treatment periods may be approved at the discretion of the Sponsor. The EAP may be discontinued at any time at the Sponsor's discretion.

At treatment discontinuation or following the end of the participant's final Treatment Period, participants will complete an end-of-study (EOS) assessment 4 weeks following discontinuation of the investigational drug product.

Visit assessments may be collected remotely, via tele-visit with study site staff. Investigational product may be shipped by the site to participants who do attend in-clinic visits.

ELIGIBILITY:
For Protocol CNMAu8.EAP01

The participants must meet the following inclusion criteria:

1. Able to understand and give written informed consent.
2. Male or female participants aged 18 years or greater (inclusive) at the time of ALS diagnosis.
3. Participants whose conditions are defined as "definite ALS" or "probable ALS" or "possible ALS" diagnostic criteria by the revised El Escorial Criteria as determined by a neurologist specializing in ALS (e.g., the Principal Investigator or sub-investigator at the site).
4. Participant is able to daily consume 60 mL of the investigational drug suspension without substantial dysphagia, OR can intake the drug through a gastrostomy tube.
5. In the judgement of the Investigator, the participant's expected survival is greater than six-months
6. Participants who have established care with a neurologist at the specialized ALS center involved in the study and will maintain this clinical care throughout the duration of the EAP.
7. Participant must have completed standard clinical safety labs within the prior 90 days from the Baseline visit including a chemistry panel (e.g., CMP) and a hematology panel (e.g., CBC).

OR Prior participation in the HEALEY Platform ALS trial (Regimen C) Open Label Extension (NCT04414345) will be considered an automatic inclusion.

Participants will be excluded from the expanded access protocol if they meet any of the following criteria:

1. Participant is eligible for a clinical study with CNM-Au8 for the treatment of ALS.
2. Participant with a history of any clinically significant or unstable medical condition based on the Investigator's judgment that may interfere with assessment of the study objectives.
3. Based on the investigator's judgment, participants who may have difficulty complying with the protocol and/or any study procedures.
4. Within the prior 90 days the participant has had clinically significant abnormalities in hematology, blood chemistry, ECG, or physical examination not resolved by the Baseline visit which according to Investigator can interfere with EAP participation.
5. Participant is currently involved in another placebo-controlled clinical trial (note: concomitant therapy with other investigational products is permitted with certain restrictions.
6. Females who are pregnant or nursing or who plan to get pregnant during the course of this EAP or within 6 months of the end of the EAP.
7. Females of child-bearing potential, or men, who are unwilling or unable to use accepted methods of birth control.
8. History of gold allergy. OR These exclusion criteria will not be applied if the participant was previously enrolled in the HEALEY Platform ALS trial (Regimen C) Open Label Extension (NCT04414345).

For Protocol CNMAu8.EAP02

Inclusion Criteria:

1. Able to understand and give written informed consent.
2. Male or female participants aged 18 years or greater (inclusive) at the time of ALS diagnosis.
3. Participants with a confirmed diagnosis of ALS per Gold Coast criteria as determined by a neurologist specializing in ALS (e.g., the site principal investigator or sub-investigator for this study).
4. Participant is able to daily consume up to 240 mL of the investigational drug suspension without substantial dysphagia, OR can intake the investigational product through a gastrostomy tube.
5. Participant must have completed standard clinical safety labs within the prior 90 days from the Baseline visit including a chemistry panel (e.g., CMP) and a hematology panel (e.g., CBC).
6. In the judgement of the Investigator the participant's expected survival is greater than six-months.
7. Participants who have established care with a neurologist at the specialized ALS center involved in the study and will maintain this clinical care throughout the duration of the EAP within the United States.

OR Prior participation in the HEALEY Platform ALS trial (Regimen C) Open Label Extension (NCT04414345) will be considered an automatic inclusion.

Exclusion Criteria:

1. Participant is eligible for participation in: (i) the HEALEY ALS Platform trial (NCT04297683), or (ii) any active study investigating CNM-Au8 for the treatment of ALS.
2. Participant has a history of any clinically significant or unstable medical condition (other than ALS) that may interfere with assessment of safety or compromise the study objectives.
3. Based on the investigator's judgment, participants who may have difficulty complying with the protocol and/or any study procedures.
4. Within the prior 90-days the participant has had clinically significant findings on standard hepatic, hematologic, or renal safety assays.
5. Participant is currently involved in another placebo-controlled clinical trial (note: concomitant therapy with other investigational products is permitted with certain restrictions.
6. Females who are pregnant or nursing or who plan to get pregnant during the EAP or within 6 months of the end of this trial.
7. Females of child-bearing potential, or men, who are unwilling or unable to use accepted methods of birth control.
8. History of gold allergy.

OR These exclusion criteria will not be applied if the participant was previously enrolled in the HEALEY Platform ALS trial (Regimen C) Open Label Extension (NCT04414345).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Barrow Neurological Institute, Phoenix, Arizona
  - UC Irvine, Orange, California
  - Sutter Health (Enrollment is full, not recruiting), San Francisco, California
  - Hospital for Special Care (Enrollment is full, not recruiting), New Britain, Connecticut
  - Nova Southeastern University, Davie, Florida
  - Northwestern (Enrollment is full, not recruiting), Chicago, Illinois
  - University of Kansas (Enrollment is full, not recruiting), Fairway, Kansas
  - Massachusetts General Hospital (Enrollment is full, not recruiting), Boston, Massachusetts
  - Henry Ford Health Systems (Enrollment is full, not recruiting), Detroit, Michigan
  - University of Nebraska Medical Center (Enrollment is full, not recruiting), Omaha, Nebraska
  - DUKE University Medical Center (Enrollment is full, not recruiting), Durham, North Carolina
  - Providence Health (Enrollment is full, not recruiting), Portland, Oregon
  - Penn State Health (Enrollment is full, not recruiting), Hershey, Pennsylvania
  - Jefferson Hospital (Enrollment is full, not recruiting), Philadelphia, Pennsylvania
  - Texas Neurology, Dallas, Texas
  - University of Washington, Seattle, Washington